CLINICAL TRIAL: NCT05759156
Title: Prophylactic Tranexamic Acid (TXA) Administration in Patients Undergoing Caesarean Delivery (CD).
Brief Title: Tranexamic Acid in Patients for Caesarian Delivery.
Acronym: TXA; CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Atif Shafqat, Assistant Professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2891
Record Dates: First submitted 2023-02-24; First posted 2023-03-08 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Postpartum Hemorrhage; Cesarean Section Complications; Obstetric Anesthesia Problems
Keywords: caesarian delivery; postpartum haemorrhage; obstetrics quality of recovery; tranexamic acid
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tranexamic Acid (Active Comparator)
  Interventions: Drug: Tranexamic acid injection
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — The intervention consists of administration of 1gm of Tranexamic acid (TXA) intravenously or 10-mls of placebo (normal saline) intravenously, slowly over 30-60 sec, within 3 mins of the delivery of baby.

SUMMARY:
This is a prospective, double-blinded, randomized placebo-controlled trial. The study will be approved by the DUHS institutional review board (IRB) and the trial will be registered at clinical trial registry. After receiving the trial information from the obstetricians during prenatal visits or from the anaesthetists during the systematic anaesthesia visit, or both the prospective women will be invited to participate in the trial. The intervention consists of administration of 1gm of tranexemic acid (TXA) or 10-mls of placebo (normal saline) intravenously, according to the randomization groups slowly over 30-60 sec, within 3 mins of the delivery of baby, after the routine prophylactic uterotonic administration and cord clamping. Administration of the prophylactic uterotonic agent (and TXA or placebo) may be followed by a two-hour oxytocin infusion, in accordance with the hospital policy. All women will be followed up at 48 hours after caeserian delivery. A venous blood sample will be obtained on day-two (D2) after delivery for outcome assessment. Adverse events will be assessed until hospital discharge and by telephone interview at 8 weeks after delivery.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria will include:

1. Informed consent of the participant
2. All women who are 18 years old or above
3. Gestational age equal or above 34 weeks
4. Women undergoing emergency or elective CD
5. Complete blood count (CBC) within seven days before the CD

Exclusion Criteria:

The exclusion criteria will include:

1. Women with thromboembolic or bleeding incidents in the past
2. Hypersensitivity to TXA
3. History of epilepsy or seizure
4. Women with abnormal placenta including accreta, increta or percreta
5. Any active cardiovascular, renal, or liver disorders
6. Autoimmune disorders
7. Sickle cell disease
8. Placenta Previa
9. Abruptio Placentae
10. Eclampsia or HELLP syndrome
11. Women who might undergo intraoperative complications.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of postpartum haemorrhage (PPH) | up to 2 days
Obstetrics quality of recovery (ObsQoR) score | at 2 days

SECONDARY OUTCOMES:
Measurement of postpartum blood loss | at 2 days
Operative time | up to 3 hours
Length of hospital stay | up to 4 days
Frequency of emergency surgery for postpartum haemorrhage | up to 12 hours
Rate of ICU transfer | up to 1 day
Rate of Maternal death | up to 3 months
Adverse events related to tranexamic acid | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- DowUHS, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No